CLINICAL TRIAL: NCT05757063
Title: Evaluation of the Effects of Two Different Sedation Protocols Used in Patients Undergoing Spinal Anesthesia on Cardiac Electrophysiology
Brief Title: Impact of Two Different Types of Sedation on ICEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Burak NALBANT, assistant professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICEB
Record Dates: First submitted 2023-02-22; First posted 2023-03-07 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Propofol; Dexmedetomidine; Electrophysiological Balance Index; QT Interval, Variation in; Tp-e Interval; QT Dispersion; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Sedation procedure with propofol
  Interventions: Other: Sedation with propofol
- Dexmedetomidine (Active Comparator): Sedation procudure with dexmedetomidine
  Interventions: Other: sedation with dexmedetomidine

INTERVENTIONS:
Other: Sedation with propofol — After spinal anesthesia, patients will be sedated with propofol.
  Arms: Propofol
Other: sedation with dexmedetomidine — After spinal anesthesia, patients will be sedated with dexmedetomidine.
  Arms: Dexmedetomidine

SUMMARY:
The QT interval is a measure of the combination of cardiac depolarization and repolarization as it encompasses both the QRS complex and the J-T interval. QT, QTc, QTd prolongation or shortening has been associated with ventricular arrhythmias . In order to define non-torsogenic drug-induced arrhythmias, the index of cardio-electrophysiological balance (iCEB), which is a new marker calculated with the QT/QRS formula, has been defined. In our study, we planned to evaluate the effects of dexmedetomidine and propofol on cardiac electrophysiology with all these parameters, especially the newly defined iCEB.

DETAILED DESCRIPTION:
Seventy patients who underwent operation under regional anesthesia and received intraoperative sedation will be included in the study. The patients will be divided into two groups, Group D (dexmedetomidine) and Group P (propofol). Sedative agent infusion will be started immediately after spinal anesthesia is administered. Preoperative ASA (American Society of Anesthesiologists) scores, demographic data, comorbidities and medications used will be recorded. Vitals and ECG prior to spinal anesthesia will be recorded. After that, spinal anesthesia will be applied and vitals and ECG will be recorded at 1, 5, 10, 15, 45 and 75 minutes. The sedation levels of the patients will be measured noninvasively by bispectral index (BIS) monitoring. Patients will be kept within the limits of light sedation. The maximum dose of 1.4 micrograms/kg/hour in the dexmedetomidine group (group D, n=35) and 4.5 milligrams/kg/hour in the propofol group (group P, n=35) will not be exceeded. The following parameters were set as the safety endpoint during sedation:

* Respiratory rate ≤8
* SpO2; 95
* Heart rate; 40
* Systolic blood pressure;80 At these endpoints, the patient's sedation dose will be reduced regardless of the BIS value.

During sedation, patients will be given 3 liters of nasal oxygen per minute, which can be increased according to need. Just before and 1st, 5th, 10th, 15th, 45th, 75th minutes after spinal anesthesia systolic arterial pressure, diastolic arterial pressure, mean arterial pressure,peak heart rate, oxygen saturation, bispectral index, QT time, QTc, QT distribution, Tpe, iCEB will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA Ⅰ-Ⅱ ,
* 18-80 years old, who will be operated under spinal anesthesia

Exclusion Criteria:

* Hypersensitivity to the propofol,dexmedotimidine
* preoperative QTc prolongation
* preoperative heart disease
* use of drugs that affect the QT interval
* severe sinus bradycardia
* preoperative electrolyte abnormalities
* liver and kidney function abnormalities
* non-sinus rhythm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
ICEBc | İntraoperative 10th minute
  QTc/QRS formula

SECONDARY OUTCOMES:
ICEB | Baseline,İntraoperative 1th,5th,10th,15th,30th,45th,75th minute
  Index of cardio-electrophysiological balance (iCEB); calculated as QT distance divided by QRS duration (QT/ QRS), it will be calculated from the ECG.
ICEBc | Baseline,İntraoperative 1th,5th,15th,30th,45th,75th minute
  QTc/QRS formula
QT | Baseline,İntraoperative 1th,5th,10th,15th,30th,45th,75th minute
  The investigator will assess the QT interval
QTc | Baseline,İntraoperative 1th,5th,10th,15th,30th,45th,75th minute
  The investigator will assess the QTc interval
QTd | Baseline,İntraoperative 1th,5th,10th,15th,30th,45th,75th minute
  maxQT-minQT
Tpe | Baseline,İntraoperative 1th,5th,10th,15th,30th,45th,75th minute
  Tpeak-Tend
Heart Rate | Baseline,İntraoperative 1th,5th,10th,15th,30th,45th,75th minute
  The investigator will assess the Heart Rate from ECG
Bispektral index | Baseline,İntraoperative 1th,5th,10th,15th,30th,45th,75th minute
  bispectral index measurement
non invaziv systolic blood pressure | Baseline,İntraoperative 1th,5th,10th,15th,30th,45th,75th minute
  non invasive systolic blood pressure measurement
non invaziv diastolic blood pressure | Baseline,İntraoperative 1th,5th,10th,15th,30th,45th,75th minute
  non invasive diastolic blood pressure measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No